CLINICAL TRIAL: NCT01372137
Title: First-in-human Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of NOX-H94
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TME Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: SNOXH94C001; 2011-000705-46 (EudraCT Number)
Record Dates: First submitted 2011-06-08; First posted 2011-06-13 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2014-06

CONDITIONS: Anemia; Chronic Diseases; Inflammation
Keywords: NOX-H94; Hepcidin; Anemia; Inflammation
MeSH Terms: conditions — Anemia; Chronic Disease; Inflammation | interventions — NOX-H94

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NOX-H94 (Experimental): Group A: single 15 minutes IV infusion of 0.3 mg/kg NOX-H94 Group B: single 15 minutes IV infusion of 0.6 mg/kg NOX-H94 Group C: single 15 minutes IV infusion of 1.2 mg/kg NOX-H94 Group D: single 15 minutes IV infusion of 2.4 mg/kg NOX-H94 Group E: single 15 minutes IV infusion of 4.8 mg/kg NOX-H94 Group F: single / repeated SC injection of NOX-H94 over a treatment period of 2 weeks Group G: multiple doses of NOX-H94 as a 15 minutes IV infusion over a treatment period of 2 weeks Group H: multiple doses of NOX-H94 as a 15 minutes IV infusion over a treatment period of 2 weeks
  Interventions: Drug: NOX-H94
- Glucose 5% (Placebo Comparator): Group A to Group H get NOX-H94 or Placebo
  Interventions: Other: Glucose 5%

INTERVENTIONS:
Drug: NOX-H94 — Dosage form: NOX-H94 25 mg (oligonucleotide basis) Solution for Injection Strength: 14.6 mg NOX-H94 / mL Dose: 0.3 - 4.8 mg/kg single dose Route: IV infusion over 15 minutes / SC administration
  Other Names: lexaptepid pegol
  Arms: NOX-H94
Other: Glucose 5% — Placebo
  Arms: Glucose 5%

SUMMARY:
This is the first clinical trial with NOX-H94. The purpose of this clinical trial is to identify a safe and efficacious treatment regimen for the clinical development of NOX-H94 in patients with anemia of chronic disease (inflammation).

DETAILED DESCRIPTION:
NOX H94 is a pegylated Spiegelmer that specifically binds to human hepcidin, thereby antagonizing its role in hemostasis, and is therefore indicated for use in anemia of inflammation. Human hepcidin has emerged as the central regulatory molecule of systemic iron homeostasis. Hepcidin expression in hepatocytes is regulated by multiple, in particular opposing signals, including systemic iron availability, hepatic iron stores, erythropoietic activity, hypoxia, and inflammatory states. These different signals are integrated transcriptionally. In chronic inflammation, such as occurs in rheumatoid arthritis, chronic kidney disease or cancer, elevated hepcidin levels have been measured and may be a key factor leading to anemia in these patients.

NOX-H94 is therefore indicated for treatment of patients with an anemia of inflammation, which is characterized by increased intracellular iron stores, increased serum ferritin concentrations and reduced sensitivity to treatment with erythropoiesis stimulating agents (ESAs), due to the limited availability of serum iron. Antagonism of hepcidin by NOX-H94 therefore leads to elevated levels of iron and transferrin saturation in the peripheral blood and could supply iron for erythropoiesis thereby correcting the anemia.

ELIGIBILITY:
Inclusion Criteria

* Male subjects or female subjects of non-childbearing potential (Groups A to E), male subjects (groups F to H)
* Age 18-65 years
* Healthy as determined by medical history, physical examination, vital signs, 12-lead electrocardiogram, and clinical laboratory parameters
* Males willing to use 2 means of contraceptive methods for at least 2 months after the final examination

Exclusion Criteria:

1. Anemia predominantly caused by other factors than chronic disease.
2. Iron overload or disturbances in utilization of iron.
3. Intravenous iron treatment or blood transfusion within 4 weeks prior to screening visit.
4. Erythropoietin treatment within 4 weeks prior to screening visit.
5. Intake of Intravenous iron, Blood transfusions, Erythropoietin during their trial participation.
6. Resting supine pulse rate < 40 or > 100 beats / min.
7. Resting supine blood pressure:

   Systolic blood pressure < 90 or > 160 mmHg Diastolic blood pressure < 40 or > 100 mmHg.
8. History or presence of confirmed orthostatic hypotension defined.
9. Positive test of HIV type 1/2 antibodies, HBs antigen, HBc antibodies, HCV antibodies.
10. Participation in another clinical trial during the last 3 months before starting this trial.
11. Positive test for drugs of abuse.
12. Diseases or condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
13. Marked repolarization abnormality.
14. Current bronchial asthma, childhood asthma which has been resolved is allowed.
15. Definite or suspected history of drug allergy or hypersensitivity or intolerance to PEG
16. Regular intake of over 14 units of alcohol per week for women and 21 units for men.
17. Not able to abstain from consumption of:

    * Caffeine containing beverages or food (tea, coffee, cola, chocolate, etc.)
    * Quinine containing beverages or food (bitter lemon, tonic water)
    * Grapefruit juice (sweet or sour)
    * Poppy seeds containing beverages or food
18. Subjects who have donated any blood, plasma or platelets in the month prior to screening
19. History of seizures or at risk
20. Known or suspected of not being able to comply with the trial protocol and/or clinical unit restrictions.
21. History of or presence of clinically significant diseases other than the underlying disease.
22. Surgery or trauma with significant blood loss within the last 2 months before administration of study drug.

28. History of increased bleeding risk.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2011-07; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | 0 to 90 days

SECONDARY OUTCOMES:
drug plasma concentrations | 0 to 29 days

CONTACTS AND LOCATIONS:
Overall Officials: Riecke Kai, MD, Study Director — TME Pharma AG
Locations (1):
- HMR, London, United Kingdom

REFERENCES:
- [Derived] Park EJ, Choi J, Lee KC, Na DH. Emerging PEGylated non-biologic drugs. Expert Opin Emerg Drugs. 2019 Jun;24(2):107-119. doi: 10.1080/14728214.2019.1604684. Epub 2019 Apr 19. PMID 30957581
- Available data/document: Manuscript: doi: 10.1111/bph.13433 — http://onlinelibrary.wiley.com/doi/10.1111/bph.13433/abstract;jsessionid=E657A6C9667BB70DE92E5B69B86B1D3F.f01t01